CLINICAL TRIAL: NCT02464618
Title: Improving Attendance to Outpatient Endoscopy Among Blacks
Brief Title: Using Patients' Social Contact to Improve Out-Patient Endoscopy Among Blacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Howard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-14-MED-11
Record Dates: First submitted 2015-06-02; First posted 2015-06-08 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-06

CONDITIONS: Compliance; Colon Cancer
Keywords: Colonoscopy; Upper endoscopy; Adherence; Disparities
MeSH Terms: conditions — Patient Compliance; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): The social contact of patients in this arm will not be contacted
- Social contact intervention (Active Comparator): The social contact of patients in this arm will be contacted and asked to facilitate the endoscopy care plan of the patient
  Interventions: Behavioral: Social contact intervention

INTERVENTIONS:
Behavioral: Social contact intervention — The social contact of the patients in this arm will be engaged to improve adherence to out-patient endoscopy
  Arms: Social contact intervention

SUMMARY:
Non-attendance to out-patient endoscopic procedures is high among underserved blacks. The overall goal of this proposal is to evaluate the effect of directly involving a social contact (chosen by the patient) on completion and quality of out-patient endoscopy recommended for the patient by his/her primary care physician, or after scheduling by the gastrointestinal endoscopist.

Improved adherence and better quality of procedures are postulated with involvement of social contacts.

DETAILED DESCRIPTION:
The overarching goal of this proposal is to determine whether directly involving a social contact, chosen by the patient, will improve the completion and quality of scheduled out-patient endoscopy among blacks.

These are three sub-projects:

Project 1: Involves recruiting 400 patients referred for colonoscopy by their primary care physicians

Project 2: Involves recruiting 400 patients scheduled for colonoscopy by their endoscopist

Project 3: Involves recruiting 200 patients scheduled for upper endoscopy by their endoscopists

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for out-patient colonoscopy by primary care physicians
* Patients scheduled for out-patient screening colonoscopy
* Patients scheduled for out-patient upper endoscopy

Exclusion Criteria:

* Patients who were referred for colorectal cancer (CRC) screening as in-patients
* Patients with personal history of familial adenomatous polyposis syndrome (FAP)
* Patients with family history of Hereditary non-polyposis colorectal cancer syndrome (HNPCC)
* Patients with inflammatory bowel disease
* Patients with Crohn's disease
* Patients with ulcerative colitis
* Patients with personal history of CRC
* Patients who have had colonic resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
Compliance with appointment and colonoscopy | 6 months
  For primary care subjects: Making appointment with Gastrointestinal endoscopist within 3 months and completing colonoscopy within 6 months of enrolment
Compliance with scheduled upper endoscopy and colonoscopy | Scheduled procedure time, an average of 8 weeks
  For specialty subjects: Completing scheduled upper endoscopy or colonoscopy

SECONDARY OUTCOMES:
Bowel preparation quality | At scheduled colonoscopy, an average of 8 weeks
  Adequacy of bowel preparation with ratings of good to excellent on Aronchick scale

OTHER OUTCOMES:
Social contact's activity | During the duration of the project, an average of 6 months
  Characteristics of participants and Lubbens social network scale correlation with other outcomes and activities of the social contact

CONTACTS AND LOCATIONS:
Overall Officials: Adeyinka O Laiyemo, MD, MPH, Principal Investigator — Howard University
Locations (1):
- Howard University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Laiyemo AO, Williams CD, Burnside C, Moghadam S, Sanasi-Bhola KD, Kwagyan J, Brim H, Ashktorab H, Scott VF, Smoot DT. Factors associated with attendance to scheduled outpatient endoscopy. Postgrad Med J. 2014 Oct;90(1068):571-5. doi: 10.1136/postgradmedj-2012-131650. Epub 2014 Sep 1. PMID 25180285
- [Background] Tammana VS, Laiyemo AO. Colorectal cancer disparities: issues, controversies and solutions. World J Gastroenterol. 2014 Jan 28;20(4):869-76. doi: 10.3748/wjg.v20.i4.869. PMID 24574761
- [Background] Badurdeen DS, Umar NA, Begum R, Sanderson AK 2nd, Jack M, Mekasha G, Kwagyan J, Smoot DT, Laiyemo AO. Timing of procedure and compliance with outpatient endoscopy among an underserved population in an inner-city tertiary institution. Ann Epidemiol. 2012 Jul;22(7):531-5. doi: 10.1016/j.annepidem.2012.04.013. Epub 2012 May 8. PMID 22571991
- [Background] Laiyemo AO. In search of a perfect solution to ensure that "no colon is left behind". Dig Dis Sci. 2012 Feb;57(2):263-5. doi: 10.1007/s10620-011-2010-6. Epub 2011 Dec 20. No abstract available. PMID 22183821
- [Derived] Laiyemo AO, Kwagyan J, Williams CD, Rogers J, Kibreab A, Jack MA, Lee EE, Brim H, Ashktorab H, Howell CD, Smoot DT, Platz EA. Using Patients' Social Network to Improve Compliance to Outpatient Screening Colonoscopy Appointments Among Blacks: A Randomized Clinical Trial. Am J Gastroenterol. 2019 Oct;114(10):1671-1677. doi: 10.14309/ajg.0000000000000387. PMID 31478919